CLINICAL TRIAL: NCT03560544
Title: Pilot Study of a Tailored Intervention to Break up Sitting in the Workplace on Cardiometabolic Risk and Worker Productivity
Brief Title: The Effect of Breaking up Sitting in the Workplace on Cardiometabolic Risk and Worker Productivity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Bedfordshire (Other)
Responsible Party: Principal Investigator, Prof David Hewson, Professor of Health and Ageing, University of Bedfordshire
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IHREC836
Record Dates: First submitted 2018-04-11; First posted 2018-06-18 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Sedentary Lifestyle
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breaking up sitting time (Experimental): A behaviour-change intervention to break up prolonged sitting in the workplace
  Interventions: Behavioral: Breaking up sitting
- Control (No Intervention): The participants in the control group will continue their daily activities as normal without any form of information about the intervention.

INTERVENTIONS:
Behavioral: Breaking up sitting — A three-part behaviour change intervention, including:
  1. Supportive organisational culture and knowledge of consequence of prolonged sitting
  2. Environmental Modification
  3. Behavioural Changes
  Arms: Breaking up sitting time

SUMMARY:
This pilot randomized controlled trial (RCT) will examine the effect of a tailored workplace intervention based on interrupting sitting on work productivity, well-being and cardio-metabolic risk in office workers. The experimental group in the 8-week intervention will be prompted to alternate between sitting and standing while working. The ratio between sitting and standing will begin at 3:1 (two hours per day in an eight-hour day) and increase to 1:1 (four hours per day in an eight-hour day) by the end of the second week of the eight-week intervention.

ELIGIBILITY:
Inclusion Criteria:

* Full-time office employees from any ethnic background, PC/Android phone users, and recruited from two different work sites.

Exclusion Criteria:

* Pregnancy
* History of musculoskeletal complaint
* Non-ambulatory
* Having a planned holiday that would mean they would not be at work for more than two weeks during the 8-week intervention period.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in sitting time (objective) | Change from baseline sitting time at 8 weeks
  Evaluation of change in sitting time in the workplace using wearable accelerometers (ActivPAL3; PAL Technologies Ltd., Glasgow, UK). The ActivPAL will be worn on the right thigh.
Change in physical activity level (objective) | Change from baseline physical activity level at 8 weeks
  Evaluation of physical activity time in the workplace using wearable accelerometers (ActivPAL3; PAL Technologies Ltd., Glasgow, UK). The ActivPAL will be worn on the right thigh.
Change in sitting time (subjective) | Change from baseline sitting time at 8 weeks
  The International Physical Activity Questionnaire (IPAQ) will be used to provide a subjective measure of sitting. The scale provides a measure of reported sitting time in minutes.
Change in physical activity level (subjective) | Change from baseline physical activity level at 8 weeks
  The International Physical Activity Questionnaire (IPAQ) will be used to provide a subjective measure of physical activity level. The scale provides a measure of reported sitting time in minutes for each of three types of physical activity (vigorous, moderate, and walking).

SECONDARY OUTCOMES:
Absenteeism | Change from baseline absenteeism at 8 weeks
  Participants will be asked to respond to questions on the Gaudine and Gregory questionnaire on unsanctioned absence. Self-reported absenteeism will be calculated by adding the number of days reported for all the three questions.
Presenteeism | Change from baseline presenteeism at 8 weeks
  Presenteeism will be measured using Work Limitations Questionnaire (WLQ). The WLQ requires employees to self-report their level of difficulty (or ability) to perform 25 specific job demands in the last 2 weeks. Answers generated for the 25 items will be grouped into four work limitation scales including Time Management; Physical Demands; Mental/Interpersonal and Output Demands. The scores for each subscale range from 0-100%, with 0 equivalent to no limitation and 100 equivalent to complete limitation.
Ecological momentary assessment (EMA) | Eight weeks
  Participants will be prompted at random four times between 9am to 5pm from Monday to Friday to complete a short questionnaire which will only take them 60 seconds to complete whilst in sitting position, standing and /or in walking position to enter their level of productivity.
Height | Once at baseline
  Measurement of height
Change in weight | Change from baseline weight at 8 weeks
  Measurement of weight
Change in waist circumference | Change from baseline waist circumference at 8 weeks
  Measurement waist circumference
Blood pressure | Change from baseline blood pressure at 8 weeks
  Systolic and diastolic blood pressure on the right arm after resting for at least 10 min in a seated position using an automated blood pressure monitor (Omron HEM705 CP, Omron Healthcare UK Limited, Milton Keynes, UK).
Change in fasting total cholesterol | Change from baseline fasting total cholesterol at 8 weeks
  Blood samples will be collected in capillary tubes after an overnight fast using a finger prick method with lancet. Measures of total cholesterol will be made.
Change in fasting high-density lipoprotein | Change from baseline fasting high-density lipoprotein at 8 weeks
  Blood samples will be collected in capillary tubes after an overnight fast using a finger prick method with lancet. Measures of high-density lipoprotein will be made.
Change in fasting triglycerides | Change from baseline fasting triglycerides at 8 weeks
  Blood samples will be collected in capillary tubes after an overnight fast using a finger prick method with lancet. Measures of triglycerides will be made.
Change in fasting blood glucose levels | Change from baseline fasting blood glucose levels at 8 weeks
  Blood samples will be collected in capillary tubes after an overnight fast using a finger prick method with lancet. Measures of blood glucose levels will be made.
Stress | Change from baseline stress at 8 weeks
  Cohen Perceived Stress questionnaire will be used to assess perception of stress. It primarily evaluates the unpredictability, uncontrollability and overload of an individual's life.
Mood | Change from baseline mood at 8 weeks
  The positive and negative affect schedule (PANAS) questionnaire is a 20-item self-report measure of both positive and negative affect.
Mental Wellbeing | Change from baseline mental wellbeing at 8 weeks
  The Warwick-Edinburgh Mental well-being Scale will be used to determine whether mental wellbeing changes. This scale has 14 questions, with each question scored from 1-5, giving a total score from 14-70.
Self-efficacy | Change from baseline self-efficacy at 8 weeks
  A generalised four-point Likert scale questionnaire will be used to measure the self-efficacy of the participants.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Bedford Borough Council, Bedford, Bedfordshire
  - University of Bedfordshire, Luton, Bedfordshire

IPD SHARING:
Plan to Share IPD: No